CLINICAL TRIAL: NCT03597165
Title: The Health Outcomes, Utility, and Costs of Returning Incidental Genomic Findings
Brief Title: Incidental Genomics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0819
Record Dates: First submitted 2018-05-31; First posted 2018-07-24 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Incidental Findings; Genomic Sequencing; Randomized Controlled Trial; Clinical Utility; Personal Utility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incidental Genomic Sequencing Results (Experimental): Patients in Intervention will receive GS results related to primary indication (cancer) and will be offered the option learning their incidental results, categorized into five "bins" based on a framework by Berg et al.
  Interventions: Other: Incidental Genomic Sequencing Results
- Primary Indication only (Active Comparator): Patients in the control will receive the intervention GS results for Primary Indications only.
  Interventions: Other: GS Results for Primary Indications only

INTERVENTIONS:
Other: Incidental Genomic Sequencing Results — Patient will receive GS results related to their primary indication (cancer), as well as the option to learn incidental GS results. Incidental results will be categorized into five "bins" based on Berg et al.'s framework (medically actionable and pharmacogenetic, common disease SNPs, Mendelian conditions, early-onset brain diseases, and carrier status). In pre-test counseling, patients will have the option to select which bins of incidental results they would like to learn, if any.
  Arms: Incidental Genomic Sequencing Results
Other: GS Results for Primary Indications only — Patients will receive GS results related to the primary indication (cancer) only.
  Arms: Primary Indication only

SUMMARY:
Health care providers (HCP) are increasingly using genomic sequencing (GS) to diagnose diseases and target treatment for patients. However, GS may incidentally reveal inherited risks for thousands of current and future diseases. Guidelines recommend HCP inform patients of incidental GS results. GS is a relatively new technology, raising many questions about its adoption in clinical care, including: What are the psychological harms, health outcomes, clinical utility and economic costs of receiving primary and incidental GS results? We will use a randomized controlled trial (RCT) to evaluate whether patients receiving incidental GS results will report higher levels of distress and more risk reducing behaviors compared to patients receiving GS for their primary indication alone. We will explore the personal utility of GS via in-depth interviews with a subset of patients. Clinical utility for cancer and incidental results will be evaluated through diagnostic yield, clinical actions triggered by GS results and in-depth interviews with a subset of patients and providers. The economic impact will be evaluated in two ways: (a) health service use will be assessed retrospectively using billing records from the Institute of Clinical Evaluative Sciences (ICES); and, (b) participants' personal costs incurred as a result of GS will be assessed via surveys. Participants will be adult cancer patients who have received negative single gene or panel test results and who have been determined by their health care provider to be a candidate for GS.

DETAILED DESCRIPTION:
Background

Genomic sequencing (GS) is considered the 'next step' towards personalized medicine, providing an opportunity to improve the prevention, diagnosis and treatment of disease. Across Canada, clinicians are increasingly using GS to identify treatments and management approaches likely to benefit patients based on molecular makeup, especially in oncology. GS offers increased sensitivity over classic genetic tests. For example, multi-gene sequencing has been shown to increase the sensitivity of identifying clinically actionable mutations in breast cancer patients by 50% to 60% when compared to testing for BRCA1/2 alone. Often breast cancer patients who test negative for BRCA1/2 will be offered GS to identify causative mutations. In addition, GS can also be used to analyze the molecular profile of a patient's tumour (somatic GS) to identify therapeutic targets.

However, the process of decoding the genome an individual or their tumour may incidentally reveal information about inherited predispositions to other cancers and diseases, including genetic variants/changes associated with current (undiagnosed) disease, drug response, risk for future diseases and variants of unknown clinical significance. Increasing policy guidance suggests that 'medically actionable' results should be offered to patients undergoing clinical sequencing, with calls to offer additional incidental results based on patient preferences. There is limited evidence on the psychological harms and clinical benefits of returning incidental GS results to patients.

Psychological distress: Single-gene and multiplex testing for hereditary cancers, neurological and cardiac disease appears to have minimal psychological impacts. A recent study found that few participants report distress from GS results. However, these findings are based on individuals who agreed to be tested for particular genes, and were prepared through counseling or otherwise to receive these results. This may not translate to incidentally-discovered genetic risk, which individuals did not anticipate or choose to learn a priori. Distress related to receiving incidental GS results remains unknown.

Personal utility: Studies suggest that individuals want to learn their GS results because they expect them to offer 'personal utility'. Personal utility is considered an increasingly important precursor of clinical utility, which is believed to offer richer self-knowledge and motivate risk reducing behaviors. Most studies focus on the hypothetical return of incidental GS results, little is known about individuals' actual perceived value of receiving GS results.

Health benefits: Single-gene and multiplex testing for low risk single nucleotide polymorphisms (SNPs) and high penetrance susceptibility alleles appears to influence the uptake of diet and medication changes, risk-reducing surgeries and surveillance. However, these findings are based on individuals who requested testing for selected genes, and may not represent individuals who learn incidental results.

Clinical Utility: Due to the challenges of applying traditional measures of clinical utility (quality adjusted life years, life years gained) in the context of genomic medicine, an 'intermediate outcome' of utility has emerged based on the 'usefulness and added value to patient management decision making,' of results captured by clinical actions or altered medical recommendations. Preliminary evidence shows GS holds great promise to enable personalized treatments and efficient diagnoses, has demonstrated to facilitate diagnosis in cases of rare diseases with unclear etiology, and strong potential to inform personalized drug therapies compatible with patients' genotypes. The utility of germline GS has largely been examined in limited clinical contexts, such as paediatrics and rare diseases. GS results have been shown to alter clinical management, such as by informing specialist referrals. In a study among a small sample of physicians, providers expressed that while they viewed the current utility of GS as low, they expect it to become more commonplace and more useful in the future. The actual and perceived utility of GS will ultimately determine its clinical implementation, and more evidence in broader clinical settings is needed to inform GS' optimal translation into clinical practice.

Economic Analysis: A lack of evidence remains around the costs and cost-effectiveness of GS. Some believe GS has potential to reduce overall healthcare spending by streamlining the diagnostic process enabling tailored treatments, and informing specific prevention efforts. Others, however, believe that GS will increase healthcare expenditures with limited clinical benefits, as sequencing and variant interpretation costs remain high and results may trigger cascades of additional testing and screening procedures. Out-of-pocket costs may be incurred by patients including medications, counseling, and peripheral costs such as lost wages and transportation. Cost-effectiveness studies have predominately been conducted in the context of tumour sequencing for pharmacological applications; the cost-effectiveness of germ-line GS for primary indication has been examined in few clinical contexts. Regarding incidental findings, cost-effectiveness studies have been conducted for fewer than one third of conditions whose disclosure is recommended by the American College of Medical Genetics and Genomics (ACMG). Modelling predicts incidental finding disclosure may be cost-effective for diagnostics but not currently for general population screening. Further investigation into the utility, costs, and cost-effectiveness of GS is necessary to inform health service delivery and funding decisions.

Rationale

It is unknown whether incidental GS results will be perceived as useful, and whether they motivate the intent or uptake of risk-reducing behaviours. The clinical utility of GS results has not been fully explored, and there is a lack of evidence around cost-effectiveness and costs associated with GS to patients and the healthcare system, which poses a barrier to its clinical implementation.

Research Question

Do patients receiving incidental GS results experience higher levels of distress and engage in more risk reducing behaviours? What is the diagnostic yield of GS, and how do GS results influence clinical decision making? What are the short-term and long-term costs associated with receiving GS results to patients and the healthcare system?

Objectives

1. Evaluate the psychological distress of receiving incidental GS results
2. Evaluate the personal utility and impact of receiving incidental GS results on subsequent risk reduction behaviours.
3. Evaluate the clinical utility of GS:

   a. Assess the diagnostic yield of GS results: i. Related to primary cancer indication. ii. Medically actionable incidental findings. iii. Incidental findings with implications for reproductive decisions, lifestyle and relatives.

   b. Explore the nature and extent of clinical activity triggered by primary and incidental GS results (referrals to specialists, laboratory testing, scans and screens, etc.).

   c. Explore patient and provider perspectives of the perceived and actual clinical utility of primary and incidental GS results.
4. Examine the short-term (1 year) and long-term (5 year) costs associated with genomic sequencing:

   1. Costs to the healthcare system.
   2. Personal costs.

Study procedures

Patients will be recruited from familial cancer clinics in the Greater Toronto Area (GTA), consented by a genetic counselor, and randomized. Following randomization, participants in the intervention arm will have the option to select which categories of incidental results they would be willing to receive, with a genetic counselor. Participants' genomes will be sequenced and interpreted. Results will be returned by a genetic counselor. Referrals will be made based on sequencing results. Outcomes will be measured at multiple time points before and after the return of results.

ELIGIBILITY:
Inclusion Criteria:

* Affected with Cancer
* Received a negative/inconclusive germline single gene test result for a cancer gene mutation (e.g., BRCA1/2, MLH, MSH, PMS, etc.) in the past two years
* Or received a negative/inconclusive germline panel test result
* 18 years old or older
* Speak and read English

Exclusion Criteria:

* Are in advanced stage cancer (stage 4 /metastatic cancer)
* Currently in active treatment (chemotherapy, radiation, scheduled surgery) - patients who are on Prophylactic Hormonal Therapy (eg tamoxifen) will be included
* Received a positive genetic test for a cancer gene mutation (e.g., BRCA1/2, MLH, MSH, PMS, APC, MUTYH, etc.)
* Have not had single gene germline testing related to their primary cancer condition (e.g., BRCA1/2 for breast/ovarian cancer, MLH, MSH, PMS colorectal cancer, etc.)
* Previously received genomic sequencing for any reason
* Currently pregnant or planning on getting pregnant (Including men whose partner is pregnant or planning). Participants who become pregnant over the course of the study will not be excluded.
* Do not speak or read English
* Under 18 years of age
* Have a family member participating in the study
* Participant in previous study of decision aid (Decision Aid RCT Study or Usability Study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 2 weeks after return of results
  Our primary outcome is distress, measured by the Hospital Anxiety & Depression Scale (HADS) using a validated cut-off of >11 on either the anxiety or depression subscale. The Hospital Anxiety and Depression Scale measures clinically significant anxiety and depression. There are two subscales, anxiety (7 items) and depression (7 items). Scores on each subscale range from 0-21, with higher scores indicating worse outcome (higher anxiety or depression). Subscale scores are not combined for a total score. (PMID: 6880820, 25005549)

SECONDARY OUTCOMES:
Impact of Event Scale-Revised (IES-R) | 1 year following return of results.
  The Impact of Event Scale-Revised (IES-R) is a standardized, validated scale that measures symptoms of traumatic stress. The IES-R comprises of three subscales: Intrusion (8 items), Avoidance (8 items), and Hyperarousal (6 items). The IES-R yields a total score that ranges from 0-88, with higher scores indicating worse outcomes. Scores on the Intrusion subscale range from 0-32, with higher scores indicating worse outcomes. Score on the Avoidance subscale range from 0-32, with higher scores indicating worse outcomes. Scores on the Hyperarousal subscale range from 0-24, with higher scores indicating worse outcomes. (PMID: 23243796)
Multi-Dimensional Impact of Cancer Risk Assessment (MICRA) | 1 year following return of results.
  The Multi-Dimensional Impact of Cancer Risk Assessment (MICRA) is a 25-item standardized, validated scale that measures the impact of result disclosure from genetic tests. There are three subscales: Distress (6 items), Uncertainty (9 items) and Positive Experiences (4 items). Total scores range from 0-125, with higher scores indicating worse outcome. Scores on the Distress subscale range from 0-30, with higher scores indicating worse outcome. Scores on the Uncertainty subscale range from 0-45, with higher scores indicating worse outcome. Scores on the Positive Experiences Subscale range from 0-20, with higher scores indicating worse outcomes. (PMID: 12433008)
Adapted Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire | 1 year following return of results.
  We will assess the intended use and actual adoption of risk-reducing behaviours and preventative services across all RCT participants using CDC's Behavioural Risk Factor Surveillance System (BRFSS) questionnaire. We have adapted the BFRSS to examine whether the receipt of GS results influences participants' intent to adopt, and actual self-reported adoption of: screening, prophylactic surgery, dietary changes, reduced alcohol intake, increased exercise, adherence/changes to medication, and smoking cessation (beyond those taken due to their cancer diagnosis). Self-reported actual or intended use of these behaviours will be ascertained over the telephone. Higher scores indicate higher uptake of health behaviours.
SF-12 | 1 year following return of results.
  The SF-12 scale measures quality of life. The SF-12 has 12 items that address physical and mental functioning. Physical and mental health composite scores range from 0 to 100, with 0 indicating the lowest possible level of health, and 100 indicating the highest possible level of health.
Genetic Self Efficacy (GSE) | 1 year following return of results.
  Consistent with the Extended Parallel Process Model (EPPM) which suggests that that higher risk results could motivate individuals to adopt risk-reducing behaviors if they perceive an increased risk of disease, as long as self-efficacy is also high, we will assess genetic self-efficacy using a standardized, validated measure (PMID: 20884465).
Risk Perception | 1 year following return of results
  Consistent with the Extended Parallel Process Model (EPPM) which suggests that that higher risk results could motivate individuals to adopt risk-reducing behaviors if they perceive an increased risk of disease, as long as self-efficacy is also high, we will assess risk perception. Participants will be asked to report their perceived likelihood of developing diseases related to their incidental results. For each disease risk, scores range from 1 to 5, and higher scores indicate higher perceived risk. (PMID: 16969872, 24131974)
Qualitative interviews with a subset of patients | 9-12 months following return of results
  We will use in-depth interviews with patients to provide further insights into the ways in which incidental results impact the quality of life and health outcomes of cancer patients receiving incidental results. Patient interviews will explore: reasons for learning incidental GS results, to whom, how and why results have been communicated, perceived utility and impact of incidental results for personal, familial or life planning.
Qualitative interviews with a subset of practitioners | 9-12 months following return of results
  Provider interviews will explore: improvements to patient management and treatment decisions on the basis of their patients' incidental results and their perceptions of the clinical, familial and personal benefits or harms of these results for patients. Interviews will also explore providers' views on any physical or physiological impacts that receipt of incidental results have had on patients.

OTHER OUTCOMES:
Perceived Utility | 1 year following return of results.
  Perceived utility of genomic sequencing results will be measured using a scale from Lupo et al. Scale values range from 0-24, with higher scores indicating higher perceived utility of genomic sequencing results. (PMID: 27019659).
Clinical actions triggered by genomic sequencing results | 1 year following return of results.
  Patient charts will be reviewed. The number and type of medical recommendations following GS will be quantified.
Impact of genomic sequencing results on reproductive behaviors | 1 year following return of results.
  Participants will be asked about whether their genomic sequencing results have impacted their reproductive decisions or reproductive planning through questions adapted from Bombard et al. (PMID: 27256091).
Decisional Conflict Scale (DCS) | 1 year following return of results.
  This standardized, validated measure will assess decisional conflict. Possible scores range from 0 to 100, with higher scores indicating higher decisional conflict (worse outcome). There are three subscales: Uncertainty, Informed, and Values Clarity. Scores on each subscale range from 0-100, with higher scores indicating worse outcome. (PMID: 7898294)
Diagnostic yield | Immediately after sequence analysis.
  Immediately after sequence analysis is complete, will record the number and frequencies of deleterious germline mutations related to the patients' phenotype over, and by subgroup: phenotype, extent of family history, transmission type, pathogenic/likely pathogenic, deleterious germline mutations known to be recurrently mutated by cancer type.
Health Information National Trends Survey (HINTS) (Adapted) | 1 year following return of results.
  An adapted version of the HINTS questionnaire will assess how participants use and access health information. (https://hints.cancer.gov/)
Economic impact of GS results | 5 years following return of results.
  Billing records held at the Institute for Clinical Evaluative Sciences (ICES) will be accessed to obtain information related to resource use following return of results, including physician visits, hospital visits, additional testing, and diagnostic tests.
Costs incurred by participants - survey questions | 1 year following return of results.
  Participants will be asked to report personal costs associated with GS results, including out-of-pocket medications as well as peripheral costs such as transportation and lost wages.
Communication of genomic sequencing results to relatives | 1 year following return of results.
  Communication of genomic sequencing results to relatives will be assessed through questions adapted from Bombard et al. that indicate which relatives they have communicated their results to (PMID: 27256091).
Cascade genetic testing among relatives | 1 year following return of results.
  Participants will be asked about which relatives, to their knowledge, have received genetic testing as a result of learning the participant's genome sequencing results.
Cascade health behaviors among relatives | 1 year following return of results.
  Participants will be asked about which relatives, to their knowledge, have changed their health behaviors as a result of the participant's genome sequencing results.
Perceptions of uncertainties in genomic sequencing (PUGS) scale | 1 year following return of results.
  This standardized, validated measure assesses perceptions of uncertainty. Scores range from 1 to 5, with higher scores indicating higher perceptions of uncertainty. (PMID: 27925165)
Tolerance of ambiguity scale | 1 year following return of results.
  This scale measures participants' tolerance of ambiguity. Scores range from 7 to 49, with higher scores indicating higher tolerance for ambiguity. (PMID: 8231339)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Bombard, PhD, Principal Investigator — St. Michael's Hospital and University of Toronto
Locations (3):
- Canada (3):
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margret Cancer Centre, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Mighton C, Reble E, Sam J, Kodida R, Shickh S, Clausen M, Hirjikaka D, Grewal S, Panchal S, Piccinin C, Aronson M, Ward T, Armel SR, Peck L, Graham T, Silberman Y, Forster N, Capo-Chichi JM, Greenfeld E, Noor A, Cohn I, Morel CF, Elser C, Eisen A, Glogowksi E, Schrader KA, Kim RH, Chan KKW, Thorpe KE, Lerner-Ellis J, Bombard Y; Incidental Genomics Study Team. Opportunistic screening for broad range of medically relevant secondary findings: Laboratory benefits and burdens. Genet Med. 2025 Oct 14:101599. doi: 10.1016/j.gim.2025.101599. Online ahead of print. PMID 41104539
- [Derived] Shickh S, Mighton C, Clausen M, Sam J, Hirjikaka D, Reble E, Graham T, Panchal S, Eisen A, Elser C, Schrader KA, Baxter NN, Laupacis A, Lerner-Ellis J, Kim RH, Bombard Y; Incidental Genomics Study Team. Clinical Utility of Genomic Sequencing for Hereditary Cancer Syndromes: An Observational Cohort Study. JCO Precis Oncol. 2024 Dec;8:e2400407. doi: 10.1200/PO-24-00407. Epub 2024 Dec 12. PMID 39666930
- [Derived] Shickh S, Clausen M, Mighton C, Gutierrez Salazar M, Zakoor KR, Kodida R, Reble E, Elser C, Eisen A, Panchal S, Aronson M, Graham T, Armel SR, Morel CF, Fattouh R, Glogowski E, Schrader KA, Hamilton JG, Offit K, Robson M, Carroll JC, Isaranuwatchai W, Kim RH, Lerner-Ellis J, Thorpe KE, Laupacis A, Bombard Y; Incidental Genomics Study Team. Health outcomes, utility and costs of returning incidental results from genomic sequencing in a Canadian cancer population: protocol for a mixed-methods randomised controlled trial. BMJ Open. 2019 Oct 7;9(10):e031092. doi: 10.1136/bmjopen-2019-031092. PMID 31594892